CLINICAL TRIAL: NCT00606827
Title: Sodium Bicarbonate Versus Saline for the Prevention of Contrast-induced Nephropathy in Patients Undergoing Coronary Angiography
Brief Title: Sodium Bicarbonate Versus Saline for the Prevention of Contrast-induced Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prato0701; POCARD0701
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Contrast-Induced Nephropathy
Keywords: Contrast-induced nephrophaty; Contrast media; Angiography; Coronary percutaneous intervention
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Bicarbonate
  Interventions: Drug: Sodium Bicarbonate
- B (Active Comparator): Saline
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Sodium Bicarbonate — Patients in the sodium bicarbonate group (154 mEq/L) received 3 ml/kg for 1 hour before contrast medium, followed by an infusion of 1 ml/kg/h for 6 hours after the procedure
  Arms: A
Drug: Isotonic Saline — Patients assigned to the isotonic saline group received 1 ml/kg/h 0.9% sodium chloride for 12 hours before and after the procedure
  Arms: B

SUMMARY:
Contrast-induced nephrophaty (CIN) accounts for more than 10% of hospital-acquired renal failure. Hydration with sodium bicarbonate is more protective than isotonic saline in animals. Limited data are available in humans. We compared the efficacy of sodium bicarbonate versus isotonic saline to prevent CIN in a large population of patients with renal dysfunction undergoing coronary angiography or intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with creatinine clearance < 60 mL/min

Exclusion Criteria:

* contrast medium administration within the previous 10 days
* end-stage renal failure requiring dialysis
* refusal to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-01; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maioli, MD, Principal Investigator — Cardiology Unit - Prato
Locations (1):
- Ospedale Misericordia e Dolce, Prato, Prato, Italy

REFERENCES:
- [Derived] Maioli M, Toso A, Leoncini M, Gallopin M, Tedeschi D, Micheletti C, Bellandi F. Sodium bicarbonate versus saline for the prevention of contrast-induced nephropathy in patients with renal dysfunction undergoing coronary angiography or intervention. J Am Coll Cardiol. 2008 Aug 19;52(8):599-604. doi: 10.1016/j.jacc.2008.05.026. PMID 18702961